CLINICAL TRIAL: NCT04753879
Title: Multi-agent Low Dose Chemotherapy (Gemcitabine, Nab-paclitaxel, Capecitabine, Cisplatin, Irinotecan) Followed by Maintenance Olaparib and Pembrolizumab in Untreated Metastatic Pancreatic Ductal Adenocarcinoma.
Brief Title: Multi-agent Low Dose Chemotherapy GAX-CI Followed by Olaparib and Pembro in Metastatic Pancreatic Ductal Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2112; IRB00267980 (Other: Johns Hopkins Medicine Institutional Review Board)
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: PARP; Gemcitabine; Nab-paclitaxel; Capecitabine; Cisplatin; Irinotecan; Olaparib; Pembrolizumab; Immunotherapy; PD-L1 (receptor blocking antibody); Anti-PD-L1; Monoclonal Antibodies; Metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Cisplatin; Irinotecan; Capecitabine; pembrolizumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nab-paclitaxel, Gemcitabine , Cisplatin, Irinotecan, Capecitabine (Experimental): Maintenance of Pembrolizumab and Olaparib
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Cisplatin; Drug: Irinotecan; Drug: Capecitabine; Drug: Pembrolizumab; Drug: Olaparib

INTERVENTIONS:
Drug: Nab-paclitaxel — 1. Patients will receive treatment Day 1 and Day 15 of each cycle (28 days).
  2. Nab-paclitaxel (80 mg/m2) will be administered IV on Day 1 and Day 15 (28 day cycle).
  3. Other Name: Abraxane
Drug: Gemcitabine — 1. Patients will receive treatment Day 1 and Day 15 of each cycle (28 days).
  2. Gemcitabine (500mg/m2) will be administered IV on Day 1 and Day 15 (28 day cycle).
  3. Other Name: Gemzar
Drug: Cisplatin — 1. Patients will receive treatment Day 1 and Day 15 of each cycle (28 days).
  2. Cisplatin (20mg/m2) will be administered IV on Day 1 and Day 15 (28 day cycle).
  3. Other Name: N/A
Drug: Irinotecan — 1. Patients will receive treatment Day 1 and Day 15 of each cycle (28 days).
  2. Irinotecan (20 mg/m2) will be administered IV on Day 1 and Day 15 (28 day cycle).
  3. Other Name: N/A
Drug: Capecitabine — 1. Patients will receive treatment Day 1-7 and Day 15-21 of each cycle (28 days).
  2. Capecitabine (500 mg) will be administered orally twice a day on days 1-7 and 15-21 of each cycle (28 days).
  3. Other Name: Xeloda
Drug: Pembrolizumab — 1. Patients will receive treatment Day 1 every other cycle (every 6 weeks) (28 days) during maintenance phase.
  2. Pembrolizumab (400 mg) will be administered IV on day 1 every other cycle (every 6 weeks).
  3. Other Name: MK-3475; Keytruda
Drug: Olaparib — 1. Patients will receive treatment on Days 1-21 during the maintenance phase.
  2. Olaparib (300 mg) will be administered orally twice a day on Days 1- 21 of each cycle (28 days).
  3. Other Name: Lynparza

SUMMARY:
The purpose of this study is to evaluate the safety and clinical activity of maintenance olaparib and pembrolizumab following multi-agent, low dose chemotherapy with gemcitabine, nab-paclitaxel, capecitabine, cisplatin, and irinotecan (GAX-CI) in patients with untreated metastatic pancreatic ductal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1 - Subject has stable disease as measured by RECIST 1.1 or iRECIST after 6 cycles of GAX-CI.
* Cohort 2 - Subject has progressive disease as measured by RECIST 1.1 and iRECIST prior to 6 cycles of GAX-CI.
* Ability to understand and willingness to sign a written informed consent document.
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Have metastatic histologically or cytologically-proven ductal pancreatic cancer.
* Patients must not have received prior treatment for pancreatic cancer.
* Have measurable disease based on RECIST 1.1.
* Willing to have to a tumor biopsy.
* Patients must have adequate organ and marrow function defined by study - specified laboratory tests.
* Woman of childbearing potential must have a negative pregnancy test and follow contraceptive guidelines as defined per protocol.
* Men must use acceptable form of birth control while on study.
* Participant understands the study regimen, its requirements, risks and discomforts, competent to report AE, understand the drug dosing schedule and use of medications to control AE.

Exclusion Criteria:

* Patients who will be considered for surgery are ineligible.
* Had chemotherapy within 5 years prior to study treatment.
* Have received any investigational drugs within 28 days prior to study treatment.
* Had surgery within 28 days of dosing of investigational agent.
* Has history of central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Require any antineoplastic therapy.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent.
* Has received prior therapy with gemcitabine, nab-paclitaxel, capecitabine, cisplatin, irinotecan, or PARP inhibitor.
* Hypersensitivity reaction to any monoclonal antibody.
* Is taking a moderate or strong CYP3A inhibitor.
* Has uncontrolled acute or chronic medical illness.
* Has known additional malignancy that is progressing and requires active treatment.
* Has received radiotherapy for pancreatic cancer.
* Have received any live vaccine or live-attenuated, any allergen hyposensitization therapy, growth factors or major surgery within 30 days prior to study treatment.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has active autoimmune disease.
* Has an active known or suspected autoimmune disease or is receiving chronic systemic steroid therapy within 7 days prior to the first dose of study drug.
* Prior tissue or organ allograft or allogeneic bone marrow transplantation.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Requirement for daily supplemental oxygen.
* Patients with a history of (non-infectious) pneumonitis/interstitial lung disease that requires steroids.
* Subject with clinically significant wound.
* Has a confirmed history of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent.
* Infection with HIV.
* Has active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or Hepatitis C virus (defined as hepatitis C virus (HCV) RNA [qualitative] is detected) infection. Patients who are Hepatitis C antibody positive and viral load negative will be permitted to enroll.
* Has uncontrolled infection.
* Unwilling to have blood drawn.
* Has known psychiatric or substance use disorder that would interfere with cooperation with the requirements of the trial.
* Woman who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) after 6 months according to RECIST 1.1 criteria. | 6 Months
  PFS is defined as the 6 month from the date of randomization to disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Progression-free Survival (PFS) after 6 months according to IRECIST criteria. | 6 months
  PFS is defined as the 6 month from the date of randomization to disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using iRECIST criteria) or death due to any cause. Per iRECIST criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.

SECONDARY OUTCOMES:
Number of participants experiencing grade 3 or above drug-related toxicities | 4 years
  • When calculating the incidence of AEs, each AE (as defined by NCI CTCAE v5.0) will be counted only once for a given subject. Estimation based on the Kaplan-Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, MD, Principal Investigator — SKCCC Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No